CLINICAL TRIAL: NCT02942966
Title: Tack Optimized Balloon Angioplasty Study for the Below The Knee Arteries Using the Tack Endovascular System®
Brief Title: Tack Optimized Balloon Angioplasty Study of the Tack Endovascular System® in Below the Knee Arteries
Acronym: TOBA II BTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA 0137
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Angioplasty; Below the Knee; PAD; Critical Limb Ischemia; Lesion; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Tack Implant (Experimental): Implantation of a Tack using the Intact Vascular Tack Endovascular System for the repair of post angioplasty dissections below the knee.
  Interventions: Device: Tack Endovascular System

INTERVENTIONS:
Device: Tack Endovascular System — Repair of post-PTA dissections using the Intact Vascular Tack Endovascular System.
  Other Names: Post-PTA Dissection Repair Implant; Tack Implant; Tack Dissection Repair Device

SUMMARY:
This is a prospective, multi-center, single-arm, non-blinded study designed to investigate the safety and efficacy of the Tack Endovascular System in the Mid/Distal Popliteal, Tibial, and Peroneal Arteries ranging in diameter from 1.5mm to 4.5mm for the treatment of post percutaneous transluminal balloon angioplasty (PTA) dissection(s) requiring repair.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females ≥ 18 years of age at the time of consent
* Female subjects of childbearing potential must have a negative pregnancy test prior to treatment and must use some form of contraception (abstinence is acceptable) through the duration of the study
* Subject has been informed of and understands the nature of the study and provides signed informed consent to participate in the study. If the subject possesses the ability to understand and provide informed consent but due to physical inability, the subject cannot sign the informed consent form (ICF), an impartial witness may sign on behalf of the subject
* Willing to comply with all required follow-up visits
* Rutherford Classification 4 or 5.
* WIfI Wound grade of 0, 1 or modified 2.
* WIfI Foot Infection grade of 0 or 1.
* Estimated life expectancy ≥1 year

Exclusion Criteria:

* Is pregnant or refuses to use contraception through the duration of the study
* Previous bypass graft in the target limb
* Acute limb ischemia, defined as symptom onset occurring less than 14 days prior to the index procedure
* Prior or planned above-ankle amputation or complete transmetatarsal amputation to the target limb (this does not apply to ray amputation of ≤2 digits, simple digital amputations or ulcer debridements)
* WIfI Foot Infection grade 2 or 3
* Any systemic infection or immunocompromised state. Patients with an ascending infection/deep foot infection or abscess/white blood count (WBC)≥12,000/or febrile state
* Endovascular or surgical procedure (not including diagnostic procedures, planned simple digital amputation or wound debridement) to the target limb less than 30 days prior to or planned for less than 30 days after the index procedure
* Existing stent implant in the target vessel
* Any other endovascular or surgical procedure (not including diagnostic procedures, planned simple digital amputation or wound debridement) less than 14 days prior to the index procedure or planned procedure less than 30 days after the index procedure
* Known coagulopathy, hypercoagulable state, bleeding diathesis, other blood disorder, or a platelet count less than 80,000/microliter or greater than 500,000/microliter
* WIfI Wound grade of 2 or 3.
* Any subject in which antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated
* Myocardial infarction, coronary thrombolysis or angina less than 30 days prior to the Index Procedure
* History of stroke or transient ischemic attack (TIA) less than 90 days prior to the Index Procedure
* Currently on dialysis
* Known hypersensitivity or contraindication to nickel-titanium alloy (Nitinol)
* Participating in another ongoing investigational clinical trial in which the subject has not completed the primary endpoint(s)
* Has other comorbidities that, in the opinion of the investigator, would preclude them from receiving this treatment and/or participating in study-required follow-up assessments
* Known hypersensitivity or allergy to contrast agents that cannot be medically managed
* Subject already enrolled into this study
* Restenotic target lesion previously treated by means other than plain balloon angioplasty and/or less than 1 year prior to index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Geraghty, MD, Principal Investigator — Washington University School of Medicine in St. Louis; George Adams, MD, Principal Investigator — Rex Hospital
Locations (49):
- United States (37):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Mission Cardiovascular Research Institute, Fremont, California
  - Denver VA Medical Center, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Amita Health Cardiovascular Associates, Elk Grove Village, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Ascension St. John Hospital, Detroit, Michigan
  - Michigan Vascular Center, Flint, Michigan
  - St. Louis Heart & Vascular, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - Novant Health Heart and Vascular Institute, Matthews, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - WakeMed Hospital, Raleigh, North Carolina
  - Lindner Research Center, Cincinnati, Ohio
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Palmetto Health USC Medical Group, Columbia, South Carolina
  - Kore Cardiovascular Research, Jackson, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Mission Research Institute, New Braunfels, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Lake Washington Vascular, PLLC, Bellevue, Washington
- Division of Angiology, Medical University Graz, Graz, Austria
- St. Anne's University Hospital Brno, Brno, Czechia
- Germany (7):
  - Karolinen-Hospital, Arnsberg
  - Franziskus-Hospital Berlin-Radiology, Berlin
  - Westküstenklinikum Heide, Heide
  - Universitätsklinikum Leipzig, Leipzig
  - Evangelisches Krankenhaus Mülheim an der Ruhr, Mülheim
  - Krankenhaus Buchholz, Nordheide
  - MEDINOS Kliniken des Landkreises Sonneberg GmbH, Sonneberg
- Hungary (2):
  - Heart & Vascular Center - Semmelweis University, Budapest
  - Bács-Kiskun County Hospital, Kecskemét
- Auckland Hospital, Auckland, New Zealand

REFERENCES:
- [Background] Conte MS, Geraghty PJ, Bradbury AW, Hevelone ND, Lipsitz SR, Moneta GL, Nehler MR, Powell RJ, Sidawy AN. Suggested objective performance goals and clinical trial design for evaluating catheter-based treatment of critical limb ischemia. J Vasc Surg. 2009 Dec;50(6):1462-73.e1-3. doi: 10.1016/j.jvs.2009.09.044. Epub 2009 Nov 7. PMID 19897335
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108
- [Derived] Adams GL, Lichtenberg M, Wissgott C, Schmidt A, Tarra T, Matricardi S, Geraghty PJ. Twenty-Four Month Results of Tack-Optimized Balloon Angioplasty Using the Tack Endovascular System in Below-the-Knee Arteries. J Endovasc Ther. 2023 Jun;30(3):393-400. doi: 10.1177/15266028221083462. Epub 2022 Mar 30. PMID 35352604
- [Derived] Geraghty PJ, Adams GL, Schmidt A, Lichtenberg M, Wissgott C, Armstrong EJ, Hertting K; TOBA II BTK investigators. Twelve-Month Results of Tack-Optimized Balloon Angioplasty Using the Tack Endovascular System in Below-the-Knee Arteries (TOBA II BTK). J Endovasc Ther. 2020 Aug;27(4):626-636. doi: 10.1177/1526602820944402. PMID 35156451

RESULTS

PARTICIPANT FLOW:
Groups:
- Tack Endovascular System (4F): Use of the Tack Endovascular System (4F) in the mid/distal popliteal, tibial and peroneal arteries ranging in diameter from 1.5mm to 4.5mm for the repair of post percutaneous transluminal balloon angioplasty (PTA) dissection(s).
Period: Overall Study
Arm/Group | Tack Endovascular System (4F)
Started | 233 (Intent to Treat (ITT) population.)
Completed | 205 (Completed 6-month follow-up)
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | Tack Endovascular System (4F)
Number analyzed (Participants) | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 157
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 39
  White | 187
  More than one race | 0
  Unknown or Not Reported | 3
BMI [Mean (Standard Deviation); unit: Kg/m^2] — Population: BMI is missing for two subjects.
  Kg/m^2
    number analyzed (Participants) | 231
    (all) | 28.8 (5.6)
BMI >= 30 [Count of Participants; unit: Participants] — Population: BMI is missing for two subjects.
  Participants
    number analyzed (Participants) | 231
    (all) | 86
ABI in treated limb [Mean (Standard Deviation); unit: ratio] — The ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery in the arm. Population: ABI information is missing for some subjects. Values ≥1.3 are censored as non-compressible.
  ratio
    number analyzed (Participants) | 198
    (all) | 0.74 (0.27)
TBI in treated limb [Mean (Standard Deviation); unit: ratio] — The ratio of systolic blood pressure measured at the toe to systolic blood pressure measured at the brachial artery. Population: TBI information is missing for some subjects
  ratio
    number analyzed (Participants) | 117
    (all) | 0.43 (0.23)
Rutherford Classification [Count of Participants; unit: Participants] — Clinical scale identifying three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss.
  Class Clinical Description
  0 Asymptomatic -no hemodynamically significant occlusive disease
  1. Mild claudication
  2. Moderate claudication
  3. Severe claudication
  4. Ischemic rest pain
  5. Minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal ischemia
  6. Major tissue loss-extending above TM level, functional foot no longer salvageable
  Participants
    0 | 0
    1 | 0
    2 | 0
    3 | 38
    4 | 78
    5 | 117
    6 | 0
Wound Grade [Count of Participants; unit: Participants] — Part of the WIfI Classification grading system created by the Society of Vascular Surgery (SVS). This system focuses on the three main factors that impact amputation risk and clinical management: Wound, Ischemia, and foot Infection (WIfI). Each of the three factors are graded on a scale from 0 to 3. The 0 represents none, 1-mild, 2-moderate and 3-severe. For the purpose of this study only, an additional Wound grade of modified 2 was added which permits some additional wounds to be included.
  Participants
    0 | 122
    1 | 91
    modified 2 | 20
    2 | 0
    3 | 0
Ischemia Grade [Count of Participants; unit: Participants] — Part of the WIfI Classification grading system created by the Society of Vascular Surgery (SVS). This system focuses on the three main factors that impact amputation risk and clinical management: Wound, Ischemia, and foot Infection (WIfI). Each of the three factors are graded on a scale from 0 to 3. The 0 represents none, 1-mild, 2-moderate and 3-severe. Population: Ischemia grade missing for some subjects
  Participants
    0: number analyzed (Participants) | 221
    0 | 115
    1: number analyzed (Participants) | 221
    1 | 55
    2: number analyzed (Participants) | 221
    2 | 28
    3: number analyzed (Participants) | 221
    3 | 23
Foot Infection Grade [Count of Participants; unit: Participants] — Part of the WIfI Classification grading system created by the Society of Vascular Surgery (SVS). This system focuses on the three main factors that impact amputation risk and clinical management: Wound, Ischemia, and foot Infection (WIfI). Each of the three factors are graded on a scale from 0 to 3. The 0 represents none, 1-mild, 2-moderate and 3-severe.
  Participants
    0 | 194
    1 | 39
    2 | 0
    3 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Number of Participants With Freedom From MALE at 6 Months and POD at 30 Days
Description: Freedom from major adverse limb events (MALE) at 6 months defined as above-ankle target limb amputation or major re-intervention to the target lesion(s) (i.e. new bypass graft, jump/interposition graft revision, or thrombectomy / thrombolysis) and perioperative death (POD) at 30 days.
Time Frame: 6 months
Population: The number of evaluable subjects for the 6 Month Primacy Efficacy Endpoint was 209.
Measure: Count of Participants; unit: Participants
Arm/Group | Tack Endovascular System (4F)
Number analyzed (Participants) | 209
Participants | 200

2. Primary Outcome: Safety - Number of Participants With MALE Plus POD at 30 Days
Description: Major adverse limb events (MALE) at 30 days defined as above-ankle target limb amputation or major re-intervention to the target lesion(s) (i.e. new bypass graft, jump/interposition graft revision, or thrombectomy / thrombolysis) and perioperative death at 30 days
Time Frame: 30 days
Population: Four subjects were not evaluable for the 30 Day primary safety endpoint due to missing the 30 day visit and no additional visits occurred beyond day 30. One subject was not evaluable for the 30 Day primary safety endpoint due to an early 30 day visit and no additional visits Day 30. These subjects were therefore not included in the denominator for the primary safety endpoint analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tack Endovascular System (4F)
Number analyzed (Participants) | 228
Participants | 3

3. Secondary Outcome: Patency - Number of Target Lesion(s) Tacked Segment(s) Patent at 6 Months
Description: Target lesion(s) tacked segment(s) patency at 6 months defined as the presence of blood flow using duplex ultrasound. If angiography is available within the 6 month follow-up visit window, it should be used in place of the duplex ultrasound. Evidence of no blood flow within the Tacked segment indicates restenosis/loss of patency.
Time Frame: 6 months
Population: Some subjects had Tack implants placed in multiple lesions
Measure: Number; unit: number of lesions
Units Other Than Participants: number of lesions
Arm/Group | Tack Endovascular System (4F)
Number analyzed (Participants) | 233
Number analyzed (number of lesions) | 303
number of lesions | 248

4. Secondary Outcome: Target Limb Salvage - Number of Participants With Freedom From Above-Ankle Target Limb Amputation at 6 Months
Description: Target Limb Salvage defined as freedom from any above-ankle target limb amputation at 6 months.
Time Frame: 6 months
Population: The number of evaluable subjects for Target Limb Salvage at 6 Months was 209.
Measure: Count of Participants; unit: Participants
Arm/Group | Tack Endovascular System (4F)
Number analyzed (Participants) | 209
Participants | 206

ADVERSE EVENTS:
Time Frame: Summary of adverse events that have been reported through 210 days
Arm/Group | Tack Endovascular System (4F)
All-Cause Mortality (participants affected / at risk) | 63/233
Serious Adverse Events (participants affected / at risk) | 179/233
Other Adverse Events (participants affected / at risk) | 137/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tack Endovascular System (4F) (N=233)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Microcytic anemia (Blood and lymphatic system disorders) | 1 (1)
Acute on chronic heart failure (Cardiac disorders) | 2 (3)
Angina at rest (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (2)
Cardiac failure aggravated (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Coronary heart disease (Cardiac disorders) | 1 (1)
Decompensated heart failure (Cardiac disorders) | 1 (1)
Decompensation cardiac (Cardiac disorders) | 3 (3)
Heart failure (Cardiac disorders) | 2 (2)
Heart failure NYHA class III (Cardiac disorders) | 1 (1)
Heart insufficiency (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
New onset angina pectoris (Cardiac disorders) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 3 (3)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Progressive angina (Cardiac disorders) | 1 (1)
Right coronary artery stenosis (Cardiac disorders) | 1 (1)
ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Coprostasis (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal hematoma (Gastrointestinal disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Ventral hernia (Gastrointestinal disorders) | 1 (1)
Acute chest pain (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Delayed healing of wound (General disorders) | 2 (2)
In-stent peripheral artery restenosis (General disorders) | 3 (3)
Opiate withdrawal symptoms (General disorders) | 1 (1)
Puncture site bleeding (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Unknown cause of death (General disorders) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1)
Cellulitis of toe (Infections and infestations) | 1 (1)
Clostridial gastroenteritis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (2)
Gangrene peripheral (Infections and infestations) | 2 (4)
Gangrene toe (Infections and infestations) | 5 (6)
Infection of amputation stump (Infections and infestations) | 1 (1)
Osteomyelitis of the foot (Infections and infestations) | 4 (5)
Phlegmon (Infections and infestations) | 1 (1)
Pneumonia, organism unspecified (Infections and infestations) | 4 (5)
Postoperative infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Spondylodiscitis (Infections and infestations) | 1 (2)
Staphylococcus aureus bacteremia (Infections and infestations) | 1 (1)
Urinary tract infection, site not specified (Infections and infestations) | 1 (1)
Wet gangrene (Infections and infestations) | 1 (1)
Abdominal wall wound (Injury, poisoning and procedural complications) | 1 (1)
Chronic subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Fracture femur (Injury, poisoning and procedural complications) | 1 (1)
Fracture of neck of femur (Injury, poisoning and procedural complications) | 1 (1)
Overdose NOS (Injury, poisoning and procedural complications) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 4 (6)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 4 (4)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Skin tear (Injury, poisoning and procedural complications) | 2 (2)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (2)
Wound bleeding (Injury, poisoning and procedural complications) | 1 (1)
Gout aggravated (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4)
Type II diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperuricemic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Prepatellar bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Basalioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Liver carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian granulosa cell tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Bleeding intracranial (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Drop attacks (Nervous system disorders) | 1 (1)
Focal epilepsy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
Syncopal attack (Nervous system disorders) | 1 (1)
TIA (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Hyperactive delirium (Psychiatric disorders) | 1 (1)
Transient psychosis (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Acute on chronic renal failure (Renal and urinary disorders) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic leg ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (2)
Digital ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Ulcer foot (Skin and subcutaneous tissue disorders) | 1 (1)
Venous ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Medical device battery replacement (Surgical and medical procedures) | 1 (1)
Abdominal aortic aneurysm (Vascular disorders) | 1 (1)
Acute limb ischemia (Vascular disorders) | 2 (2)
Anterior tibial artery perforation (Vascular disorders) | 1 (1)
Arterial occlusion (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Atherosclerosis of arteries of the extremities (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 8 (10)
Critical limb ischemia (Vascular disorders) | 3 (3)
Digital necrosis (Vascular disorders) | 1 (1)
Dry gangrene foot (Vascular disorders) | 1 (2)
Dry gangrene toe (Vascular disorders) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Internal hemorrhage (Vascular disorders) | 1 (1)
Ischemic limb pain (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease Fontaine stage IV (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease aggravated (Vascular disorders) | 4 (5)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 9 (10)
Peripheral vascular disease (Vascular disorders) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (1)
Superficial femoral artery occlusion (Vascular disorders) | 1 (1)
Uncontrolled hypertension (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tack Endovascular System (4F) (N=233)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Microcytic anemia (Blood and lymphatic system disorders) | 1 (1)
Acute on chronic heart failure (Cardiac disorders) | 2 (3)
Angina at rest (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (2)
Cardiac failure aggravated (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Coronary heart disease (Cardiac disorders) | 1 (1)
Decompensated heart failure (Cardiac disorders) | 1 (1)
Decompensation cardiac (Cardiac disorders) | 3 (3)
Heart failure (Cardiac disorders) | 2 (2)
Heart failure NYHA class III (Cardiac disorders) | 1 (1)
Heart insufficiency (Cardiac disorders) | 2 (2)
Ischaemic heart disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
New onset angina pectoris (Cardiac disorders) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 3 (3)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Progressive angina (Cardiac disorders) | 1 (1)
Right coronary artery stenosis (Cardiac disorders) | 1 (1)
ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Meniere's disease aggravated (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Coprostasis (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2)
Melena (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal hematoma (Gastrointestinal disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Ventral hernia (Gastrointestinal disorders) | 1 (1)
Acute chest pain (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Delayed healing of wound (General disorders) | 3 (3)
In-stent peripheral artery restenosis (General disorders) | 3 (3)
Leg edema (General disorders) | 2 (2)
Opiate withdrawal symptoms (General disorders) | 1 (1)
Puncture site bleeding (General disorders) | 1 (1)
Swelling of limb (General disorders) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1)
Cellulitis of toe (Infections and infestations) | 1 (1)
Clostridial gastroenteritis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (2)
Gangrene peripheral (Infections and infestations) | 3 (5)
Gangrene toe (Infections and infestations) | 5 (6)
Infection of amputation stump (Infections and infestations) | 1 (1)
Osteomyelitis of the foot (Infections and infestations) | 4 (5)
Phlegmon (Infections and infestations) | 1 (1)
Pneumonia, organism unspecified (Infections and infestations) | 4 (5)
Postoperative infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Spondylodiscitis (Infections and infestations) | 1 (2)
Staphylococcus aureus bacteremia (Infections and infestations) | 1 (1)
Urinary tract infection, site not specified (Infections and infestations) | 1 (1)
Vascular access site infection (Infections and infestations) | 1 (1)
Wet gangrene (Infections and infestations) | 1 (1)
Abdominal wall wound (Injury, poisoning and procedural complications) | 1 (1)
Chronic subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Fracture femur (Injury, poisoning and procedural complications) | 1 (1)
Fracture of neck of femur (Injury, poisoning and procedural complications) | 1 (1)
Overdose NOS (Injury, poisoning and procedural complications) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 8 (10)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 9 (10)
Post procedural bleeding (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 4 (4)
Post procedural hematoma (Injury, poisoning and procedural complications) | 3 (3)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5)
Skin tear (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 3 (4)
Wound bleeding (Injury, poisoning and procedural complications) | 1 (1)
Gout aggravated (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4)
Type II diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperuricemic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain of lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Prepatellar bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Basalioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Liver carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian granulosa cell tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Bleeding intracranial (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Drop attacks (Nervous system disorders) | 1 (1)
Focal epilepsy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
Syncopal attack (Nervous system disorders) | 1 (1)
TIA (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Hyperactive delirium (Psychiatric disorders) | 1 (1)
Transient psychosis (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Acute on chronic renal failure (Renal and urinary disorders) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic leg ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (2)
Digital ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Ulcer foot (Skin and subcutaneous tissue disorders) | 1 (1)
Venous ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Medical device battery replacement (Surgical and medical procedures) | 1 (1)
Abdominal aortic aneurysm (Vascular disorders) | 1 (1)
Acute limb ischemia (Vascular disorders) | 2 (2)
Anterior tibial artery perforation (Vascular disorders) | 1 (1)
Arterial occlusion (Vascular disorders) | 1 (1)
Arterial spasm (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 2 (2)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Artery dissection (Vascular disorders) | 1 (1)
Atherosclerosis of arteries of the extremities (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 8 (10)
Critical limb ischemia (Vascular disorders) | 3 (3)
Deep vein thrombosis leg (Vascular disorders) | 1 (1)
Digital necrosis (Vascular disorders) | 3 (3)
Dry gangrene foot (Vascular disorders) | 1 (2)
Dry gangrene toe (Vascular disorders) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Internal hemorrhage (Vascular disorders) | 1 (1)
Ischemic limb pain (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease Fontaine stage IV (Surgical and medical procedures) | 1 (1)
Peripheral arterial occlusive disease aggravated (Vascular disorders) | 5 (6)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 9 (10)
Popliteal artery occlusion (Vascular disorders) | 1 (1)
Reperfusion injury (Vascular disorders) | 2 (2)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (1)
Superficial femoral artery occlusion (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
Tibial artery occlusion (Vascular disorders) | 1 (1)
Tibial artery stenosis (Vascular disorders) | 1 (1)
Tibial artery thrombosis (Vascular disorders) | 1 (1)
Uncontrolled hypertension (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI acknowledges that Clinical Trial is part of multi-center clinical study. Publication of multi-center data requires prior review and consent of both Sponsor and all participating sites. PI agrees that the first publication of the results of the Clinical Trial shall be made in conjunction with results from other participating sites. Provided, however, that if no multi-center publication is made within one year from database lock, then PI may publish individually.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT02942966/Prot_SAP_000.pdf